CLINICAL TRIAL: NCT02282215
Title: An Open-Label Phase 2 Prospective, Randomized, Controlled Study of CLT-008 Myeloid Progenitor Cells as a Supportive Care Measure During Induction Chemotherapy for Acute Myeloid Leukemia
Brief Title: Safety and Efficacy of Human Myeloid Progenitor Cells (CLT-008) During Chemotherapy for Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellerant Therapeutics (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CLT008-03
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Acute Myeloid Leukemia; Neutropenia; Infection
Keywords: Fever; Induction chemotherapy; Infection; Leukemia; Myeloid progenitor cells; Neutropenia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neutropenia; Infections; Fever; Leukemia | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CLT-008 low dose with G-CSF (Experimental): Dose escalation
  Interventions: Biological: CLT-008; Biological: G-CSF
- CLT-008 high dose with G-CSF (Experimental): Dose escalation
  Interventions: Biological: CLT-008; Biological: G-CSF
- CLT-008 with G-CSF (Experimental): Randomized
  Interventions: Biological: CLT-008; Biological: G-CSF
- G-CSF (Active Comparator): Randomized
  Interventions: Biological: G-CSF

INTERVENTIONS:
Biological: CLT-008 — Single intravenous infusion
  Other Names: human allogeneic myeloid progenitor cells (hMPC); romyelocel-L
  Arms: CLT-008 high dose with G-CSF; CLT-008 low dose with G-CSF; CLT-008 with G-CSF
Biological: G-CSF — Daily subcutaneous injections
  Other Names: Neupogen (filgrastim); granulocyte colony-stimulating factor; Zarxio; Granix (tbo-filgrastim)

SUMMARY:
The purpose of the study is to explore the safety and efficacy of CLT-008 as an extra supportive care measure after induction chemotherapy for patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
The prolonged period of severe neutropenia caused by induction chemotherapy for the treatment of AML is associated with a nearly universal risk of febrile neutropenia. Standard supportive care strategies include administration of prophylactic anti-bacterial and anti-fungal agents, but serious breakthrough bacterial and fungal infections still occur. Granulocyte colony-stimulating factor (G-CSF; filgrastim, Neupogen®) has been shown to shorten the duration of severe neutropenia, fever, antibiotic use and hospitalization following induction chemotherapy for AML. CLT-008, a human allogeneic myeloid progenitor cell product, is intended to provide the cellular target for G-CSF to produce neutrophils during the period of chemotherapy-induced bone marrow suppression when the patient's own progenitor cells may be limited in responding to G-CSF. It is hypothesized that the production of allogeneic neutrophils from CLT-008 will be sufficient to mitigate the infection-related consequences of induction chemotherapy for AML.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia arising de novo (per European LeukemiaNet)
2. Treated with any established chemotherapy regimen based on either:

   1. 7+3: Standard-dose cytarabine 100-200 mg per meter squared continuous infusion for 7 days with idarubicin 12 mg per meter squared or daunorubicin 45-90 mg per meter squared for 3 days
   2. High-dose cytarabine-based (HIDAC) chemotherapy administering a total cytarabine dose of ≥ 4 g per meter squared alone or in combination with other anti-leukemic agents (for example, anthracyclines, purine nucleoside inhibitors, etoposide, etc.)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at Screening or by the day chemotherapy is initiated
4. Adequate respiratory function with a room air oxygen saturation of at least 92%
5. Adequate cardiac function defined as an ejection fraction of at least 45%
6. Serum bilirubin ≤ 1.5 times the upper limits of normal. Subjects with a history of Gilbert's syndrome may be enrolled if the total bilirubin is < 3 mg/dL with an indirect bilirubin of > 1.5 mg/dL
7. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times upper limits of normal prior to chemotherapy
8. Serum creatinine ≤ 2 times upper limits of normal or estimated glomerular filtration rate ≥ 60 mL/min/1.73 meter squared per Modification of Diet in Renal Disease equation (MDRD)
9. All subjects, except post-menopausal women, must be willing to utilize a highly effective method of contraception throughout the study
10. Adequately informed of the nature and risks of the study with written informed consent

Exclusion Criteria:

1. Pregnant or breast feeding
2. Overt central nervous system manifestations of leukemia at diagnosis
3. Specifically diagnosed and uncontrolled fungal, bacterial, viral, or other infection (e.g. confirmed sepsis, pneumonia, abscess, cellulitis, etc.) at the day chemotherapy is initiated. "Uncontrolled" is defined as exhibiting ongoing signs and symptoms of infection without improvement despite antimicrobial or other treatment.
4. AML subtype M3 (promyelocytic leukemia)
5. Previous chemotherapy for AML
6. History of or current human immunodeficiency virus (HIV) or hepatitis C virus infection
7. History of or current clinically significant immunodeficiency
8. Known contraindication to receiving G-CSF
9. History of or current clinically significant alloimmunization to leukocyte antigens
10. Participation in another clinical study within 28 days of the day chemotherapy is initiated, in which the study drug or device may influence hematopoiesis. Co-enrollment in another study is allowed in cases where the investigational therapy under study is a version of an acceptable chemotherapy regimen for this study per the inclusion criteria.
11. Receiving any agent concurrently with CLT-008 infusion which inhibits cell division (e.g., methotrexate or hydroxyurea)
12. Acute or chronic medical disorder that, in the opinion of the investigator or medical monitor, may prevent the subject from completing participation in the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Duration of febrile episodes (fever) | 42 days

SECONDARY OUTCOMES:
Time to absolute neutrophil count (ANC) recovery | 42 days
Incidence and duration of febrile neutropenia | 42 days
Incidence and duration of infection | 42 days
Incidence and severity of mucositis | 42 days
Incidence of infusion reactions | 42 days
Incidence of Graft-versus-Host Disease (GVHD) | 42 days
Incidence of Adverse Events (AE) | 42 days
Incidence of Serious Adverse Events (SAE) | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: William Reed, MD, Study Director — Cellerant Therapeutics
Locations (22):
- United States (22):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation Clinic, Indianapolis, Indiana
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - University of Minnesota Physicians BMT Clinic, Minneapolis, Minnesota
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Desai PM, Brown J, Gill S, Solh MM, Akard LP, Hsu JW, Ustun C, Andreadis C, Frankfurt O, Foran JM, Lister J, Schiller GJ, Wieduwilt MJ, Pagel JM, Stiff PJ, Liu D, Khan I, Stock W, Kambhampati S, Tallman MS, Morris L, Edwards J, Pusic I, Kantarjian HM, Mamelok R, Wong A, Van Syoc R, Kellerman L, Panuganti S, Mandalam R, Abboud CN, Ravandi F. Open-Label Phase II Prospective, Randomized, Controlled Study of Romyelocel-L Myeloid Progenitor Cells to Reduce Infection During Induction Chemotherapy for Acute Myeloid Leukemia. J Clin Oncol. 2021 Oct 10;39(29):3261-3272. doi: 10.1200/JCO.20.01739. Epub 2021 Jun 22. PMID 34156898
- See also: Cellerant Therapeutics CLT-008: Myeloid Progenitor Cells — http://www.cellerant.com/pipeline/clt-008-myeloid-progenitor-cells.html